CLINICAL TRIAL: NCT01295736
Title: Evaluation of the Efficacy of Sildenafil on Time to Healing in Patients With Scleroderma and Ischaemic Digital Ulcers: a Prospective, Longitudinal, Randomized, Comparative, Double-blind, 2-parallel-arm, Placebo-controlled Study
Brief Title: Sildenafil Effect on Digital Ulcer Healing in sClerodErma SEDUCE STUDY
Acronym: SEDUCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-021135-13; 2010_14 (Other: sponsor)
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2012-07

CONDITIONS: Systemic Scleroderma
Keywords: scleroderma; digital; ulcer
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Ulcer | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Actif arm (Active Comparator): Sildenafil 20mg TID during 90 days
  Interventions: Drug: Sildenafil
- Sugar pill (Placebo Comparator): Placebo pills TID during 90 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil 20 mg TID per os during 90 days
  Arms: Actif arm
Drug: placebo — Placebo pills TID per os during 90 days
  Arms: Sugar pill

SUMMARY:
Digital ulcers (DUs) are an expression of the microangiopathy in patients with scleroderma (SSc). DUs lead to pain and impaired hand use. DUs remain a severe complication for many patients and effective therapy remains elusive. In the present study, the investigators propose to evaluate the efficacy of Sildenafil in DUs healing in a randomized double blind control study in SSc patients.

DETAILED DESCRIPTION:
This is a multicenter, prospective, longitudinal, randomized, comparative, double-blind, 2-parallel-arm, placebo-controlled study aimed to evaluate the efficacy of sildenafil 20 mg TID study on time to healing of DUs in SSc patients with ischaemic DUs.

Approximately 120 patients aged from 18 years and above will be allocated to receive either placebo or sildenafil 20mg TID during 90 days. All potential subjects will present with ischaemic digital ulcers complicating scleroderma. An eligible digital ulcer must be beyond the proximal interphalangeal joint, on finger surface (included periungual ulcers), of ischemic origin according to the physician, and not over subcutaneous calcifications or bone relief.

ELIGIBILITY:
Inclusion Criteria:

* Patient with systemic sclerosis (ScS) according to the classification criteria of the American College of Rheumatology or of "LeRoy" and "Medsger".
* ScS patient with at least one ongoing ischaemic hand digital ulcer at baseline (see below the eligibility conditions of a digital ulcer).
* Patient must have provided written informed consent prior to enrolment. Patient agrees to come to the follow up visits inside the protocol specified range.
* Relative to each DU: DU must be beyond the proximal interphalangeal joint, on finger surface, of ischemic origin according to the physician, and not over subcutaneous calcifications or bone relief.

Exclusion Criteria:

* PAH requiring PDE5 inhibitors or prostacyclin history of stroke, myocardial infarction or life threatening arrhythmia within the last 6 months
* severe cardiac failure (NYHA IV) or unstable angina within the last 6 months.
* hereditary degenerative retinal disorders non-arteritic anterior ischemic optic neuropathy or untreated proliferative diabetic retinopathy
* uncontrolled diabetes mellitus
* Patient with known severe lung obstructive disease (FEV1<70% on last available pulmonary function tests).
* severe hepatic impairment
* Patient with known impairment of renal function (serum creatinine > 2.5 ULN).
* Patient with severe malabsorption or any severe organ failure (e.g., lung, kidney) or any life-threatening condition.
* Patient who has had surgical sympathectomy performed in the previous 12 months.
* Patient with a history of upper extremity deep vein thrombosis or lymphedema within the previous 3 months.
* Patient participating in a clinical trial or having participated in a clinical trial within the previous 3 months.
* Patient having received a treatment with sildenafil for digital ulcers or pulmonary arterial hypertension within 3 months prior to inclusion.
* Patient having received a treatment with parenteral prostanoids (prostaglandin E, epoprostenol, treprostinil sodium or other prostacyclin analogs) within 3 months prior to inclusion.
* Patient having received a treatment with inhaled or oral prostanoids one month prior to inclusion.
* Patient with previous intolerance or allergy to PDE5 inhibitors or a history of multiple clinically significant allergies.
* Pregnant or lactating female.
* Patient with uncontrolled tachyarrhythmias or bradyarrhythmias, or placement of pacemaker or implantable defibrillator within 60 days prior to randomization.
* Patient with hemodynamic instability or systolic arterial pressure less than 90 mmHg and/or symptomatic orthostatic hypotension.
* Patient receiving all forms of prostacyclin or nitrates or nitric oxide donors in any form including Nicorandil.
* Patient receiving potent inhibitors of CYP3A4 such as ketoconazole, itraconazole, ritonavir.
* Patient with any condition that prevents compliance with the protocol or adhering to therapy.
* Patient who has donated blood during the previous month or intends to donate blood or blood products during the study or for one month following completion of the study.
* Patient under guardianship (including curators) or deprived of liberty.
* Patient presenting with an anatomic malformation of penis (such as an angulation, sclerosis of erectile tissue or "Lapeyronie's disease").
* Patient presenting with a disease which predisposes to priapism (such as sickle-cell disease, myeloma or leukemia).
* Patient presenting with at least one digital ulcer meeting the exclusion criteria (see below).
* Relative to each DU:
* Digital ulcer due to conditions other than scleroderma.
* Non ischaemic digital ulcer.
* Infected digital ulcer requiring systemic antibiotherapy.
* Digital ulcer requiring urgent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
time to healing of ischemic digital ulcers (DUs) in patients with scleroderma treated by sildenafil 20 mg TID versus placebo for 90 days | 90 days

SECONDARY OUTCOMES:
To evaluate the time to healing of ischemic DUs (2 mm at entry and > 1 month and <3 months old) in patients with scleroderma treated by sildenafil 20 mg TID versus placebo for 90 days. | 90 days
To evaluate the change in the number of ischaemic DUs between baseline and day 90. | 90 days
To evaluate the proportion of patients with complete healing of all DUs present at baseline at day 90. | 90 days
To evaluate the proportion of patients with complete healing of all DUs (baseline DUs and new DUs) at day 90. | 90 days
To evaluate the proportion of patients who do not develop any new DU after 28 days of treatment with the study drug up to day 90. | 90 days
To evaluate the change between baseline and day 90 in hand function and pain. | 90 days
To evaluate the proportion of patients with complicated DUs (infection, gangrene, amputation, DU requiring IV prostanoids) over the 90 days period of treatment. | 90 days
To evaluate the evolution of the severity of Raynaud's phenomenon between baseline and day 90. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric HACHULLA, PU-PH, Principal Investigator — University Hospital, Lille
Locations (24):
- France (24):
  - University Hospital, Nice, Nice, Alpes-Maritimes
  - Hautepierre Hospital, Strasbourg, Bas-Rhin
  - Nord Hospital, Marseille, Bouches du Rhone
  - CHU de Caen, Caen, Calvados
  - CHU Dijon, Dijon, Côte d'Or
  - CHU Dupuytren / dermatology, Limoges, Haute Vienne
  - CHU Dupuytren / Médecine Interne, Limoges, Haute Vienne
  - CHU de Rennes, Rennes, Ile Et Vilaine
  - University Hospital, Tours, Tours, Indre-et-Loire
  - University Hospital, Grenoble, Grenoble, Isère
  - University Hospital, Nantes, Nantes, Loire-Atlantique
  - CHU de Reims, Reims, Marne
  - University Hospital, Fort de France, Fort de France, Martinique
  - University Hospital, Lille, Lille, Nord
  - St Louis Hospital, Paris, Paris
  - University Hospital, Rouen, Rouen, Seine-Maritime
  - University Hospital, Amiens, Amiens, Somme
  - Hôpital Edouard Herriot, Lyon
  - Jean Verdier Hospital, Bondy, Île-de-France Region
  - La Pitié - Salpétriêre Hospital, Paris, Île-de-France Region
  - Cochin Hospital / Médecine Interne, Paris, Île-de-France Region
  - Cochin Hospital, Paris, Île-de-France Region
  - Saint Antoine Hospital, Paris, Île-de-France Region
  - Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region

REFERENCES:
- [Derived] Hachulla E, Hatron PY, Carpentier P, Agard C, Chatelus E, Jego P, Mouthon L, Queyrel V, Fauchais AL, Michon-Pasturel U, Jaussaud R, Mathian A, Granel B, Diot E, Farge-Bancel D, Mekinian A, Avouac J, Desmurs-Clavel H, Clerson P; SEDUCE study group. Efficacy of sildenafil on ischaemic digital ulcer healing in systemic sclerosis: the placebo-controlled SEDUCE study. Ann Rheum Dis. 2016 Jun;75(6):1009-15. doi: 10.1136/annrheumdis-2014-207001. Epub 2015 May 20. PMID 25995322